CLINICAL TRIAL: NCT00995670
Title: Ischemia/Reperfusion Injury of Human Endothelium: Role of Glucose and Statins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CARA-023-09S
Record Dates: First submitted 2009-10-13; First posted 2009-10-15 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Hyperglycemia
Keywords: hyperglycemia; statin; blood vessels; ischemic preconditioning; Anesthesia, inhalational; endothelium; 5% dextrose
MeSH Terms: conditions — Hyperglycemia | interventions — Glucose; Ascorbic Acid; Simvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sevoflurane and Glucose (Experimental): Endothelial function will be measured via forearm blood flow (FBF). Subjects may get I/R injury (ischemia) without glucose or sevoflurane (placebo); I/R with glucose only (glucose trial); I/R with sevoflurane only (sevo trial); I/R with glucose and sevoflurane (combo trial). Baseline FBF was taken in every trial before any intervention, and FBF was taken during intervention and post I/R.
  Glucose: 5% dextrose will be infused at 12 ml/hr to a target of 200 mg/dl blood concentration in the experimental forearm for 1 hr to prevent the anesthetic preconditioning (sevoflurane) protection against subsequent I/R injury.
  Sevoflurane: 1 minimum alveolar concentration (MAC) for 20 min (after 1 hr glucose and before I/R) 26 volunteers were studied 67 times in this arm.
  Interventions: Drug: 5% dextrose; Drug: Sevoflurane
- Vitamin C and Glucose (Experimental): To determine if vitamin C can restore the impairment of the endothelium (FBF) caused by the glucose (dextrose infusion). All subjects received glucose and I/R injury (ischemia), either with or without vitamin C. Control baseline FBF was taken in every trial before any intervention, and FBF was taken during intervention and post I/R.
  Placebo data were the placebo studies from the Sevoflurane and Glucose arm, when appropriate; new subjects (not enrolled in Sevoflurane and Glucose arm) underwent a separate placebo trial.
  Glucose: 5% dextrose will be infused at 12ml/hr to a target of 200 mg/dl blood concentration in the experimental forearm for 60 min.
  Vitamin C: 1 gm iv bolus injection 5 min before I/R injury 16 volunteers were studied 25 times in this arm.
  Interventions: Drug: 5% dextrose; Drug: Vitamin C
- Statins and Glucose (Experimental): Volunteers ingested a 40 mg simvastatin (statin) pill for the two evenings prior to study day and the morning of the study to determine the effect of simvastatin on modulating the I/R injury during hyperglycemia (high glucose). Volunteers were studied with statin alone and with statin and glucose.
  Placebo data were the placebo studies from the Sevoflurane and Glucose arm, when appropriate; new subjects (not enrolled in Sevoflurane and Glucose arm) underwent a separate placebo trial.
  Glucose: 5% dextrose will be infused at 12ml/hr to a target of 200 mg/dl blood concentration in the experimental forearm for 60 min.
  Statin: 40 mg of simvastatin 17 volunteers were studied 31 times in this arm.
  Interventions: Drug: 5% dextrose; Drug: Simvastatin

INTERVENTIONS:
Drug: 5% dextrose — Glucose is infused to prevent the anesthetic preconditioning (sevoflurane) protection against subsequent ischemia/reperfusion injury.
  Other Names: Glucose
Drug: Vitamin C — Vitamin C is intended to restore the impairment of the endothelium caused by the dextrose infusion.
  Other Names: Vit C
  Arms: Vitamin C and Glucose
Drug: Simvastatin — Simvastatin will be ingested to determine the efficacy of a statin to modulate the forearm response to glucose.
  Other Names: Statin
  Arms: Statins and Glucose
Drug: Sevoflurane — Sevoflurane will be given to attenuate or prevent the I/R injury during glucose.
  Other Names: Sevo
  Arms: Sevoflurane and Glucose

SUMMARY:
Anesthetic preconditioning (APC, a brief exposure to an anesthetic gas) has become an area of intense research interest because of its ability to protect tissue and organs from injury resulting from a cessation of blood flow and then a re-establishment of flow. The blood vessel lining plays a key role in this injury. This research will examine, in human volunteers, several important modifiers of APC in human blood vessels: high blood sugar, vitamin C, and statin drugs. Thus, the proposed studies will advance the investigators' understanding of mechanisms of this injury in humans and explore important modifiers of APC protection from injury.

DETAILED DESCRIPTION:
Injury to vital organs and tissue can occur when blood flow is stopped and then re-established. This happens in a variety of clinical situations and contributes to poor outcomes. A newer concept of protection from this injury by an anesthetic drug might occur because of the effect of the volatile anesthetics on the tissue that lines blood vessels. Thus, a brief exposure to a volatile anesthetic before a cessation of blood flow, called anesthetic preconditioning (APC), can substantially reduce the resulting injury to the lining of the blood vessels. In animal models, high levels of blood sugar block this protection, while cholesterol lowering drugs (statins) restore the protection and may independently protect blood vessel lining from injury. The interactions of high blood sugar and statin drugs on the blood vessel reaction to APC and a subsequent 20-min cessation of blood flow to the forearm will be studied in humans. In addition, the involvement of reactive oxygen species (ROS) in the harmful effects of high blood sugar and the beneficial effects of statins will be explored. The following four hypotheses will be studied: 1) high blood sugar blocks the anesthetic protection of blood vessels from injury in a dose and time dependent manner; 2) reactive oxygen species are involved in the inhibition of APC by high blood sugar; 3) statins modulate injury in a dose related manner; and 4) statins reduce high blood sugar inhibition of APC.

A standard model to evaluate forearm blood vessel function will be used. Thin rubber-band-like strain gauges will be strapped around each forearm and the change in their stretch during a variety of interventions on the experimental arm (the other arm will not receive any interventions and will be the control arm) will be measured. These interventions will allow the investigator to determine whether the hypotheses listed above are true. During all studies, there will be a 20-min arrest of the forearm circulation. Additional effects of injury, APC, high blood sugar, and statins will be determined by evaluating blood vessel inflammatory responses from "markers" in blood samples taken before and after I/R injury. Several studies will involve varying the forearm blood glucose concentration for brief (30 min) to longer (2 hours) periods prior to APC and injury. The ROS scavenger vitamin C will be used to evaluate the role of ROS in adverse effects of high blood sugar. There are several other studies that will continue to seek the mechanism of action of this effect via the use of other drug interactions.

ELIGIBILITY:
Inclusion Criteria:

* Young, healthy volunteers, 18-35 yr of age;
* Females will be studied at the same phase of their estrous cycle in each protocol.

Exclusion Criteria:

* Beta-blocker therapy or any medication that might interfere with vascular responses;
* Pregnant or lactating women;
* Substance abusers;
* Smokers;
* Anyone with cardiovascular, renal, or other systemic disease including hypertension and/or diabetes;
* Also excluded are volunteers with family history of malignant hyperthermia, or significant gastro-esophageal reflux.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2010-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Ebert, MD PhD, Principal Investigator — Zablocki VA Medical Center, Milwaukee
Locations (1):
- Zablocki VA Medical Center, Milwaukee, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers were sought from our research subject database.
Pre-assignment Details: None. This was not a clinical intervention study but basic science research in young healthy humans. Primary exclusion criteria included anyone on beta-blockers or other med that would affect vascular responses; pregnant or lactating women; substance abusers; smokers; and cardiovascular, renal or systemic disease including hypertension & diabetes.
Groups:
- Sevoflurane and Glucose: Endothelial function will be measured via forearm blood flow (FBF). Subjects may get I/R injury (ischemia) without glucose or sevoflurane (placebo trial); I/R with glucose only (glucose trial); I/R with sevoflurane only (sevoflurane trial); I/R with glucose and sevoflurane (combined trial). Control baseline FBF was taken in every trial before any intervention, and FBF was taken during intervention and post I/R.
- Vitamin C and Glucose: To determine if vitamin C can restore the impairment of the endothelium (FBF) caused by the glucose (dextrose infusion). All subjects received glucose and I/R injury (ischemia), either with or without vitamin C. Control baseline FBF was taken in every trial before any intervention, and FBF was taken during intervention and post I/R.
- Statin and Glucose: Volunteers ingested a 40 mg simvastatin (statin) pill for the two evenings prior to study day and the morning of the study to determine the effect of simvastatin on modulating the I/R injury during hyperglycemia (high glucose). Volunteers were studied with statin alone and with statin and glucose.
Period: Overall Study
Arm/Group | Sevoflurane and Glucose | Vitamin C and Glucose | Statin and Glucose
Started | 26 | 16 | 17
Completed | 25 (These 26 subjects underwent a total of 58 studies to determine the effect of dose of glucose on I/R.) | 16 (These 16 subjects underwent a total of 25 studies on the effect of Vitamin C.) | 14 (These 17 volunteers underwent 33 studies on the effect of statins, glucose, and glucose & statins.)
Not Completed | 1 | 0 | 3
Not completed — Failed arterial cannulation | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Population: All volunteers served as their own controls (placebo) and participated in one or more interventions, after each of which the study was repeated.
Groups:
- Sevoflurane and Glucose: Endothelial function will be measured via forearm blood flow (FBF). Subjects may get I/R injury (ischemia) without glucose or sevoflurane (placebo trial); I/R with glucose only (glucose trial); I/R with sevoflurane only (sevoflurane trial); I/R with glucose and sevoflurane (combined trial). Control baseline FBF was taken in every trial before any intervention, and FBF was taken during intervention and post I/R.
  Glucose: 5% dextrose will be infused at 12ml/hr to a target of 200 mg/dl blood concentration in the experimental forearm for 60 min to prevent the anesthetic preconditioning (sevoflurane) protection against subsequent I/R injury.
  Sevoflurane: 1 minimum alveolar concentration (MAC) for 20 min (after hour of glucose and before I/R) 26 volunteers were studied 67 times in this arm.
- Statin and Glucose: Volunteers ingested a 40 mg simvastatin (statin) pill for the two evenings prior to study day and the morning of the study to determine the effect of simvastatin on modulating the I/R injury during hyperglycemia (high glucose). Volunteers were studied with statin alone and with statin and glucose.
  Placebo data were the placebo studies from the Sevoflurane and Glucose arm, when appropriate; new subjects (not enrolled in Sevoflurane and Glucose arm) underwent a separate placebo trial.
  Glucose: 5% dextrose will be infused at 12ml/hr to a target of 200 mg/dl blood concentration in the experimental forearm for 60 min.
  Statin: 40 mg of simvastatin 17 volunteers were studied 31 times in this arm.
- Total: Total of all reporting groups
Arm/Group | Sevoflurane and Glucose | Vitamin C and Glucose | Statin and Glucose | Total
Number analyzed (Participants) | 26 | 16 | 17 | 59
Age, Customized [Number; unit: participants] — Age range of participants was 18 to 35 years of age.
  participants
    18-35 years old | 26 | 16 | 17 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 9 | 33
  Male | 12 | 6 | 8 | 26
Region of Enrollment [Number; unit: participants]
  United States | 26 | 16 | 17 | 59

OUTCOME MEASURES:

1. Primary Outcome: Forearm Blood Flow
Description: endothelial (forearm blood flow) responses to acetylcholine stimulation at baseline, and under conditions of high glucose before and after ischemia/reperfusion injury, and same with the addition of an intervention: sevoflurane (Arm 1), vitamin C (Arm 2), and high statin (Arm 3).
Time Frame: Baseline, Glucose Control, 15-min post ischemia
Measure: Mean (Standard Error); unit: ml/100 ml tissue/min
Groups:
- Sevoflurane and Glucose: To determine the effectiveness of anesthetic preconditioning (APC) via sevoflurane to attenuate the I/R injury during the normal glucose state and during hyperglycemia.
- Vitamin C and Glucose: To determine if vitamin C can restore the impairment of the endothelium caused by the dextrose infusion.
- Statin and Glucose: To determine the effect of simvastatin on modulating the I/R injury during the normal glucose state and during hyperglycemia.
Arm/Group | Sevoflurane and Glucose | Vitamin C and Glucose | Statin and Glucose
Number analyzed (Participants) | 26 | 16 | 17
ml/100 ml tissue/min
  Baseline | 6.48 (0.86) | 9.2 (2.92) | 7.32 (1.06)
  Control, Glucose | 8.26 (1.00) | 9.2 (2.92) | 9.91 (1.43)
  Post Ischemia, Glucose | 7.10 (0.65) | 7.6 (2.42) | 7.00 (1.01)
  Intervention Baseline | 8.47 (0.82) | 8.84 (1.39) | 8.17 (1.06)
  Control, after intervention | 7.90 (0.84) | 9.3 (1.73) | 9.28 (1.34)
  Post Ischemia, intervention | 8.45 (1.18) | 9.91 (1.63) | 6.26 (0.82)

ADVERSE EVENTS:
Groups:
- Sevoflurane & Glucose: To determine the effectiveness of anesthetic preconditioning (APC) via sevoflurane to attenuate the I/R injury during the normal glucose state and during hyperglycemia.
- Vitamin C & Glucose: To determine if vitamin C can restore the impairment of the endothelium caused by the dextrose infusion.
- Statins & Glucose: To determine the effect of simvastatin on modulating the I/R injury during the normal glucose state and during hyperglycemia.
Arm/Group | Sevoflurane & Glucose | Vitamin C & Glucose | Statins & Glucose
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/26 | 0/16 | 0/17

LIMITATIONS AND CAVEATS:
Some substudies were not completed because we had difficulty creating ischemia/reperfusion (I/R) injury or a consistent FBF response, which was critical to the purpose of the study to investigate the role of glucose and statins in I/R injury.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes